CLINICAL TRIAL: NCT05633472
Title: The Roles of Vitamin D and Microbiome in Children With Post-acute COVID-19 Syndromes (PACS) and Long COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH111-REC2-122
Record Dates: First submitted 2022-11-30; First posted 2022-12-01 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Post-acute COVID-19 Syndromes
Keywords: Post-acute COVID-19 Syndromes (PACS); Long COVID; human microbiome; vitamin D
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Treatment group (Experimental): Vitamin D (2000IU/day) for 6 months
  Interventions: Other: Vitamin D
- Placebo Comparator: Control group (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vitamin D — Vitamin D (2000IU/day) for 6 months
  Arms: Experimental: Treatment group
Other: Placebo — Placebo
  Arms: Placebo Comparator: Control group

SUMMARY:
A double-blind study to evaluate the role of human microbiome and vitamin D in the development of long COVID and PACS in children.

DETAILED DESCRIPTION:
Children worldwide are at risk of SARS-CoV-2 infection because of a lack of approved vaccines for children aged 0-4 years. Moreover, SARS-CoV-2 infected children also suffered with long term sequels of virus infection, which involved multiple organs, such as fatigue, post-exercise malaise, skeletal muscular pains, headache, palpitation and insomnia. In fact, there is limited evidence available on the long-term impact of SARS-CoV-2 infection in children. Recent studies have shown critical-ill COVID-19 patients suffered with low vitamin D concentration and microbiome dysbiosis in their respiratory and gastrointestinal system. Vitamin D has been known to counteract several respiratory virus infections as well as beneficial functions in multiple organs. Also, commensal microbiota in lung and intestinal tracts exert protective functions against virus infections and, through its metabolite and axis links, has anti-inflammatory actions and homeostasis in multiple organs. Hence, in this study, the investigators hypothesis that long COVID or post-acute COVID syndrome (PACS) in children is due to the effect of post-virus infection on the immuno-metabolism change (vitamin D deficiency) and perturbation of gut microbiota (microbiome dysbiosis), therefore our study aims are first, make the comparisons of vitamin D levels and respiratory and gut microbiome between symptomatic and non-symptomatic post-COVID children using cross-sectional study. Next, for interventional study, patients will be divided in two groups to receive supplementation of vitamin D or placebo for 6 months to evaluate the effect of vitamin D on the symptoms relieve and improvement of microbiome dysbiosis in post-acute COVID syndrome (PACS) children. The investigators expect through this study, the investigators can learn more on the pathogenesis and the effect of vitamin D and microbiota in long COVID and PACS in children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 0-18 years
2. The child sought/needed primary or secondary medical care for COVID-19
3. Laboratory (RT-PCR, COVID-19 antigen tests or SARS-CoV-2 antibody testing) or physician confirmed SARS-CoV-2 infection based on classic clinical symptoms and/or ground-glass opacification on CT imaging.
4. 28 days - 3 months from the onset of COVID-19 symptoms
5. Parent's/carer's/guardians consent to participate

Exclusion Criteria:

1. Recruit patients who have used antibiotics, systemic steroids, and immunosuppressants in the previous month.
2. Patients with C1 esterase inhibitor deficiency, lymphocytopenia, thrombocytopenia, severe diseases involving heart, liver, or kidney, metabolic disease, or autoimmune disease.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Levels of vitamin D | Month 0
  Vitamin D will be measured in a blood sample by ELISA to determine baseline status.
Levels of vitamin D | Month 6
  Vitamin D will be measured in a blood sample to follow the change from baseline in vitamin D level at month 6.
Single nucleotide polymorphism of vitamin D receptor and vitamin D binding protein | Month 0
  Single nucleotide polymorphism (SNP) genotyping will be performed in a blood sample by using TaqMan SNP genotyping assays.
Microbiome | Month 0
  Nasal and anal swabs will be used to detect respiratory and intestinal microbiome by using 16S rRNA sequencing to determine baseline status.
Microbiome | Month 6
  Nasal and anal swabs will be used to detect respiratory and intestinal microbiome by using 16S rRNA sequencing,and to follow the change from baseline in microbiome at month 6.
Total immunoglobulin E (IgE) | Month 0
  Plasma total IgE concentration will be measured by microparticle immunoassay (IMx analyzer, Abbott Laboratories, Abbott Park, IL) and ELISA to determine baseline status.
Total immunoglobulin E (IgE) | Month 6
  Plasma total IgE concentration will be measured by microparticle immunoassay (IMx analyzer, Abbott Laboratories, Abbott Park, IL) and ELISA to follow the change from baseline in total IgE at month 6.
Allergen-specific immunoglobulin E (IgE) | Month 0
  Plasma allergen-specific IgE will be measured by BioIC ®.

SECONDARY OUTCOMES:
Children's Somatic Symptoms Inventory (CSSI) | Month 0 to Month 6
  CSSI. Range (0-4); lower scores indicate better health
KINDL questionnaire | Month 0 to Month 6
  For assessing Health-Related Quality of Life in children and adolescents aged 3 years and older.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan